CLINICAL TRIAL: NCT06171178
Title: A Phase 1, Open-Label, Dose Escalation and Expansion Study of ASP1012, an Oncolytic Virus, in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of ASP1012 in Adults With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to strategic decision made by the sponsor the study was terminated
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1012-CL-0101
Record Dates: First submitted 2023-12-07; First posted 2023-12-14 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor
Keywords: Locally Advanced Solid Tumors; Metastatic Solid Tumors; ASP1012; Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: ASP1012 Dose Escalation (Experimental): Participants with previously treated solid tumor types will receive ASP1012 in a 21-day cycle.
  Interventions: Drug: ASP1012
- Part 2: ASP1012 Dose Expansion (Monotherapy) (Experimental): Participants with previously treated melanoma will receive ASP1012 with dose level(s) selected from dose escalation (Part 1) in a 21-day cycle.
  Interventions: Drug: ASP1012
- Part 2: ASP1012 + Pembrolizumab Dose Expansion (previously treated solid tumors) (Experimental): Participants with previously treated solid tumors, will receive ASP1012 in a 21-day cycle. Pembrolizumab will also be administered every three weeks in a 21-day cycle, for up to 3 doses.
  Interventions: Drug: ASP1012; Drug: Pembrolizumab
- Part 2: ASP1012 + Pembrolizumab Dose Expansion (treatment-naïve melanoma) (Experimental): Participants with treatment-naïve melanoma will receive ASP1012 in a 21-day cycle. Pembrolizumab will also be administered every three weeks in a 21-day cycle, for up to 3 doses.
  Interventions: Drug: ASP1012; Drug: Pembrolizumab
- Part 3: ASP1012 Dose Expansion (previously treated gastric cancer) (Experimental): Participants with previously treated gastric cancer will receive ASP1012 with dose level selected from dose escalation (Part 1) in a 21-day cycle.
  Interventions: Drug: ASP1012
- Part 3: ASP1012 Dose Expansion (colorectal cancer [CRC]) (Experimental): Participants with CRC will receive ASP1012 with dose level selected from dose escalation (Part 1) in a 21-day cycle.
  Interventions: Drug: ASP1012
- Part 3: ASP1012 Dose Expansion (ovarian cancer) (Experimental): Participants with ovarian cancer will receive ASP1012 with dose level selected from dose escalation (Part 1) in a 21-day cycle.
  Interventions: Drug: ASP1012
- Part 3: ASP1012 Dose Expansion (other solid tumor type) (Experimental): Participants with other solid tumor type will receive ASP1012 with dose level selected from dose escalation (Part 1) in a 21-day cycle.
  Interventions: Drug: ASP1012

INTERVENTIONS:
Drug: ASP1012 — Intravenous (IV) infusion
Drug: Pembrolizumab — IV infusion
  Arms: Part 2: ASP1012 + Pembrolizumab Dose Expansion (previously treated solid tumors); Part 2: ASP1012 + Pembrolizumab Dose Expansion (treatment-naïve melanoma)

SUMMARY:
ASP1012 is a type of virus called an oncolytic virus which is used to treat some cancers.

ASP1012 was changed in a laboratory to infect and kill cancer cells, leaving healthy cells alone. It also makes the cancer cells visible to the immune system which will fight the cancer cells.

Before ASP1012 is available as a treatment, the researchers need to understand how it is processed by and acts upon the body. This will help find a suitable dose for future studies and check for potential medical problems from the treatment.

In this study, ASP1012 is being tested in humans for the first time. ASP1012 has already been tested in the laboratory and in animals. This is the standard way new potential treatments are developed.

People in this study will be adults whose tumor has either grown outside of the area where it started (locally advanced) or it has spread to other parts of the body (metastatic). They will receive ASP1012. Also, some people will receive ASP1012 with pembrolizumab, an approved medicine.

There are 2 main aims of this study. The first is to learn if people with certain solid tumors can tolerate different doses of ASP1012. The second is to find a suitable dose of ASP1012.

This study will be in 3 parts.

Part 1 is called Dose Escalation. People with locally advanced or metastatic tumors can take part. They will have been previously treated with all available standard cancer therapies. Different small groups of people will receive lower to higher doses of ASP1012.

For each dose, any medical problems will be recorded. This will help to find suitable doses of ASP1012 to use in Parts 2 and 3 of the study. The first group will receive the lowest dose of ASP1012. A medical expert panel will check the results from this group and decide if the next group can receive a higher dose of ASP1012. The panel will do this for each group until all groups have taken ASP1012 or until suitable doses have been selected for Parts 2 and 3.

Part 2 is called Dose Expansion. 3 groups will take part: people with previously-treated melanoma (a type of skin cancer) that have not responded to their treatment (refractory) or their cancer has come back (relapsed), people with newly-diagnosed or untreated melanoma, and people with previously-treated solid tumors. People with previously-treated melanoma will receive ASP1012 at the dose worked out from Part 1. People with previously-treated solid tumors will receive ASP1012 with pembrolizumab. The first few people will receive ASP1012 at a lower dose than the dose worked out from Part 1, to check the safety of the treatments being given together. If there are no safety issues: the next people in the solid tumor group will receive ASP1012 at the dose worked out from Part 1, with pembrolizumab; also people with untreated melanoma will receive ASP1012 at the dose worked out from Part

1, with pembrolizumab.

Part 3 is also a Dose Expansion for people with other specific cancers. These are stomach cancer, ovarian cancer, or colorectal cancer. If people with certain tumors respond well in Parts 1 and 2 of the study, other people with this same type of tumor can also take part in Part 3.

For all parts of the study, ASP1012 will be given through a vein. This is called an infusion.

Each treatment cycle is 21 days long. People will start with 3 treatment cycles. People in the study may receive extra treatment cycles, if they respond well to treatment. People with melanoma who are receiving ASP1012 with pembrolizumab will not be offered the extra treatment cycles. People can stop leave the study early if: they have medical problems from the treatment; their cancer gets worse; they start other cancer treatment; they ask to stop treatment; or they do not come back for treatment.

People will visit the clinic on certain days during their treatment. Some visits will be virtual or by phone. During all clinic visits, the study doctors will check for any medical problems from ASP1012. They will also check vital signs. Vital signs include temperature, pulse, breathing rate, the amount of oxygen in the blood, and blood pressure. At some visits, other checks will also include a medical examination, and an electrocardiogram (ECG) to check the heart rhythm, blood draws and urine samples for testing. A tumor sample, if available, will be taken during the first treatment cycle. People will have imaging scans and have blood draws for testing every 6 weeks during and after treatment. This will stop if they leave the study early.

People will visit the clinic within 7 days and 30 days after stopping treatment. At both visits, the study doctors will check for any medical problems from ASP1012. Other checks will include a medical examination, blood draws and urine samples for testing and checking vital signs. An ECG will also be done at the 7-day visit. After the 30-day visit, clinic staff will phone people in the study every 12 weeks to check the condition of their cancer for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Parts 1 and 2 must have histologically, or cytologically, confirmed diagnosis of locally advanced or metastatic solid tumor(s).

  * Dose Escalation (Part 1) - all previously treated participants with solid tumor types
  * Dose Expansion (Part 2)
  * Participants with previously treated cutaneous melanoma, that is, anti-programmed cell death protein 1 (PD-1)/programmed death ligand 1 (PD-L1) alone or in combination with anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitor. Participants with BRAF-mutant melanoma must have received a v-raf murine sarcoma viral oncogene homolog B (BRAF) inhibitor as monotherapy or in combination with other targeted agents (for example, murine embryonic fibroblasts (MEK) inhibitors).
  * Participants with previously treated solid tumors,
  * Participants with stage IIIB to IIID or oligometastatic resectable stage IV, treatment-naïve melanoma that are amenable to resection.

Note: Participants with acral lentiginous melanoma will be excluded.

* Participants in Part 3 (Dose Expansion) must have histologically, or cytologically confirmed diagnosis of either:

  * Previously treated (at least 1 line of prior therapy) gastric cancer (including gastroesophageal junction cancer [type 2 and 3 only]). Prior lines of therapy may include combination chemotherapy such as FOLFOX based regimen containing 5-flurouracil, leucovorin and oxaliplatin, targeted therapies against human epidermal growth factor receptor 2 (HER2+) tumors and checkpoint inhibitors.
  * Stage II to IV CRC in complete remission with no measurable disease as defined by RECIST v1.1 following surgical resection and adjuvant therapy with circulating tumor deoxyribonucleic acid (ctDNA) detectable by local testing; the ctDNA positivity will be confirmed during the trial by centralized testing Note: Participants with Stage IV CRC are limited to those with oligometastatic disease in liver. Participants with CRC must have received and completed standard of care and adjuvant therapies which may include fluoropyrimidine, oxaliplatin, bevacizumab, and irinotecan-based chemotherapy and surgery.
  * Stage II to IV ovarian cancer including breast cancer gene mutations in complete remission with no measurable disease as defined by RECIST v1.1 following surgical resection and adjuvant therapy with CA-125 concentration exceeding 2 times of normal level (> 70 units per milliliter [U/mL]) as measured by local testing. Participants with ovarian cancer must have received standard of care and adjuvant therapies which may include platinum-based chemotherapy and/or poly-ADP ribose polymerase (PARP) inhibitors.
  * Other solid tumor type (when identified), for example, a tumor type in which antitumor activity or biomarker response is observed in Parts 1 or 2 or additional tumor types of interest.
* Participant has measurable disease as determined by RECIST v1.1, except for participants with CRC and ovarian cancer enrolled in Part 3. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participant has progressed, relapsed or discontinued for toxicity during or after the last systemic anti-neoplastic therapy and is unlikely to achieve clinical benefit from standard of care therapies per investigator, except for Part 2 participants with treatment-naïve melanoma and Part 3 (participants with CRC and ovarian cancer). There is no limit to the number of prior anti-neoplastic therapies received.
* Participant has a predicted life expectancy ≥ 12 weeks.
* Participant has at least 1 site of disease suitable for biopsy (except for Part 3 [participants with CRC and ovarian cancer]) and is willing and able to undergo required tumor biopsies according to the treating institution's guidelines at screening and during study treatment. Bone biopsies are not acceptable.
* Participant has an ECOG performance status of 0 or 1.
* Female participant:

  * Is not pregnant and at least 1 of the following conditions apply:
  * Not a woman of child bearing potential (WOCBP)
  * WOCBP who has a negative urine or serum pregnancy test at screening and agrees to follow the contraceptive guidance from the time of informed consent throughout the treatment period and for at least 180 days after the final ASP1012 administration.
  * Must not be breastfeeding or lactating starting at screening and throughout the treatment period and 180 days after the final ASP1012 administration.
  * Must not donate ova starting at first administration of study intervention and throughout the treatment period and for 180 days after the final ASP1012 administration.
* Male participant:

  * Must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 180 days after the final ASP1012 administration.
  * Must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 180 days after the final ASP1012 administration.
  * Must not donate sperm during the treatment period and for 180 days after the final ASP1012 administration.
* Participant must be willing and able to comply with the study requirements including prohibited concomitant medication restrictions.
* Participant agrees not to participate in another interventional study while receiving ASP1012 in the present study/participating in the present study.

Exclusion Criteria:

* Participant has ongoing toxicity ≥ Grade 2 per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 considered clinically significant and attributable to prior anti-neoplastic therapies. Note: Participants with peripheral neuropathy, type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy or skin disorders (for example, vitiligo, psoriasis, or alopecia) not requiring systemic treatment are allowed.
* Participant has had major surgery ≤ 4 weeks of signing the informed consent form (ICF).
* Participant has symptomatic or untreated central nervous system metastases or leptomeningeal disease. Participants with treated symptomatic brain metastases should be neurologically stable (for 4 weeks post-treatment and prior to screening) and off steroids for at least 2 weeks prior to first administration of ASP1012.
* Participant has active or prior autoimmune or inflammatory disorders requiring systemic therapy within the past 2 years (including inflammatory skin conditions, or inflammatory bowel disease [for example, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], celiac disease, systemic lupus erythematosus, non-infectious pneumonitis, Sarcoidosis syndrome, Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis). The following are exceptions to this criterion:

  * Participant with type 1 diabetes mellitus
  * Participant with vitiligo or alopecia
  * Participant with endocrinopathies stably maintained on appropriate replacement therapy.
  * Participant with any chronic skin condition that does not require systemic therapy
* Participant with eczema or history of eczema requiring systemic treatment.
* Participant with another malignancy that currently requires treatment
* Participant with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of first administration of ASP1012. Inhaled or topical steroids and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Participant has received a prior allogeneic bone marrow or solid organ transplant.
* Participant has a condition requiring use of anti-viral agents with a potential to inhibit vaccinia replication. Prophylactic use of anti-viral agents (e.g., acyclovir) is permitted.
* Participant has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, any form of substance abuse or psychiatric illness/social situations that would limit compliance with study visits or requirements or a condition that could invalidate communication.
* Participant has a known history of human immunodeficiency virus (HIV) infection or suffers from other acquired and congenital immunodeficiency diseases. HIV testing is not required for the purposes of this study unless mandated by local health authority.
* Participant has a history of moderate to severe ascites, clinically significant and/or rapidly accumulating ascites, bleeding esophageal varices, hepatic encephalopathy or pericardial and/or pleural effusions related to liver insufficiency.
* Participant has a clinically significant abnormal ECG at screening that imposes a safety risk for participation in the study.
* Participant has symptomatic cardiovascular disease within the preceding 12 months including but not limited to the following: significant coronary artery disease (for example, requiring angioplasty or stenting), acute myocardial infarction or unstable angina pectoris < 3 months prior to screening, uncontrolled hypertension, clinically significant arrhythmia or congestive heart failure (New York Heart Association grade ≥ 2), pericarditis or myocarditis < 3 months prior to screening.

Prior/Concomitant Therapy

* Participant has received a live vaccine against infectious diseases or COVID-19 vaccine within 28 days prior to the first dose of ASP1012. If a participant has received Paxlovid for COVID-19, a 1-week washout period is required prior to the first dose of ASP1012.
* Participant has received prior radiation therapy within 2 weeks of the first dose of ASP1012. Participant must have recovered from all radiation-related toxicities, not require corticosteroids and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system disease.

Prior/Concurrent Clinical Study Experience

* Participant is concurrently participating in another interventional study or has received an investigational product or other immunotherapy anti-cancer therapy or anti-viral therapy ≤ 30 days or 5 half-lives, whichever is shorter, prior to first administration of ASP1012.

Diagnostic Assessments

* Participant with inadequate organ and marrow functions meeting any of the below criteria:

  * Leukocytes < 3000/microliter (µL)
  * Absolute neutrophil count < 1500/µL (for participants with known Duffy null or benign ethnic neutropenia, absolute neutrophil count < 1000/μL)
  * Platelets < 100 000/µL
  * Hemoglobin < 9 grams per deciliter (g/dL)
  * International normalized ratio (INR) > 1.5 × upper limit of normal (ULN) and/or activated partial thromboplastin time > 1.5 × institutional normal limits total bilirubin (TBL) > 1.5 × institutional normal limits (participants with known Gilbert syndrome who are excluded if TBL > 3.0 × institutional normal limits or direct bilirubin > 1.5 × institutional normal limits) aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3.0 × institutional normal limits; Participants with tumors in the liver, AST and/or ALT > 5 × institutional normal limits
  * Albumin < 2.5 g/dL
  * Creatinine clearance < 45 milliliter per minute (mL/min) (calculated by Cockcroft-Gault equation). Alternatively, GFR < 45 mL/min/1.73 m^2 (calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation) can be used.
* Participant has any of the following per screening serology test:

  * Hepatitis A virus antibodies (immunoglobulin M)
  * Positive hepatitis B surface antigen (HBsAg) or detectable hepatitis B virus (HBV) DNA. Participants with negative HBsAg, positive hepatitis B core antigen and negative hepatitis B surface antibodies are eligible if HBV DNA is undetectable.
  * HCV antibodies unless hepatitis C virus (HCV) ribonucleic acid (RNA) is undetectable
* Positive coronavirus 2019 antigen test 10 days prior to cycle 1 day 1 (C1D1) with ASP1012

Other Exclusion Criteria

* Participant has any condition, which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP1012 or any components of the formulation used, including prior adverse reaction to vaccinia (for example, as smallpox vaccine).
* Participant has had previous exposure with ASP1012 or known exposure (< 5 years) to pox virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Up to 28 days
  A DLT will be defined as any event meeting the DLT criteria occurring during the DLT assessment period that is considered possibly, probably or definitely related to ASP1012.
Number of participants with Adverse Events (AEs) | Up to 19 months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Note: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the (study) procedures.
Number of participants with laboratory value abnormalities and/or AEs | Up to 7 months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to 7 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 6 months
  Number of participants with potentially clinically significant ECG values.
Number of participants at each grade of Eastern Cooperative Oncology Group (ECOG) performance status scores | Up to 7 months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.

SECONDARY OUTCOMES:
ASP1012 viral DNA in blood | Up to 7 months
  Viral DNA will be measured by quantitative polymerase chain reaction (qPCR) to ascertain viral load.
Viral shedding of ASP1012 in urine | Up to 7 months
  Viral DNA will be analyzed by qPCR and plaque assay.
Viral shedding of ASP1012 in saliva | Up to 7 months
  Viral DNA will be analyzed by qPCR and plaque assay.
Viral shedding of ASP1012 in feces (part 1) | Up to 6 months
  Viral DNA will be analyzed by qPCR and plaque assay.
Number of participants with positive anti-drug antibodies to ASP1012 | Up to 6 months
Objective Response Rate (ORR) per Immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to 19 months
  ORR is defined as the proportion of participants whose best overall response is a confirmed Complete Response (CR) or Partial Response (PR).
ORR per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 19 months
  ORR is defined as the proportion of participants whose best overall response is a confirmed Complete Response (CR) or Partial Response (PR).
Duration of Response (DOR) per iRECIST | Up to 19 months
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented progressive disease (PD) or death due to any cause, whichever occurs first.
DOR per RECIST v1.1 | Up to 19 months
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented PD or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) per iRECIST | Up to 19 months
  DCR is defined as the proportion of participants whose best overall response is rated as confirmed CR, PR or stable disease.
DCR per RECIST v1.1 | Up to 19 months
  DCR is defined as the proportion of participants whose best overall response is rated as confirmed CR, PR or stable disease.
Overall Survival (OS) | Up to 19 months
  OS is defined as the time from the start of study treatment to date of death due to any cause.
Progression Free Survival (PFS)/ Relapse Free Survival (RFS) per iRECIST | Up to 19 months
  PFS/RFS is defined as the time from the start of study intervention to first documentation of PD or death due to any cause, whichever comes first.
PFS/RFS per RECIST v1.1 | Up to 19 months
  PFS/RFS is defined as the time from the start of study intervention to first documentation of PD or death due to any cause, whichever comes first.
Major Pathologic Response (MPR) | Up to 19 months
  MPR is defined as the proportion of participants whose pathologic response is rated as pathological complete response (pCR) or near pCR.
Amount of viral DNA in tumor tissues | Up to 19 months
  The viral genomic load will be quantified using a validated qPCR assay in tumor tissue samples.
Change from baseline in cancer antigen 125 (CA-125) (Ovarian cancer only) | Baseline to month 19
  Change from baseline will be summarized with descriptive statistics.
Change from baseline in circulating tumor DNA (ctDNA) (CRC only) | Baseline to month 19
  Change from baseline will be summarized with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development, Inc.
Locations (8):
- United States (8):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa Hospitals, Iowa City, Iowa
  - Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Gabrail Cancer and Research Center, Canton, Ohio
  - Mary Crowley Cancer Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/